CLINICAL TRIAL: NCT05408390
Title: Effects of Energy and Physical Density Manipulation on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: US Army Research and Development Command- Soldier Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 22-03HC; M-10975 (Other: US Army Medical Research and Development Command IRB)
Record Dates: First submitted 2022-05-24; First posted 2022-06-07 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Appetite; Eating Behavior
Keywords: Appetite; Eating behavior; Energy density
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low physical and energy density (Experimental)
  Interventions: Other: LPD+LED
- High physical and low energy density (Experimental)
  Interventions: Other: HPD+LED
- Low physical and high energy density (Experimental)
  Interventions: Other: LPD+HED
- High physical and energy density (Experimental)
  Interventions: Other: HPD+HED

INTERVENTIONS:
Other: LPD+LED — Low physical density (LPD) + low energy density (LED) foods. Participants receive breakfast, lunch and snack items engineered to have LPD and LED.
  Arms: Low physical and energy density
Other: HPD+LED — High physical density (HPD) + low energy density (LED) foods. Participants receive breakfast, lunch and snack items engineered to have HPD and LED.
  Arms: High physical and low energy density
Other: LPD+HED — Low physical density (LPD) + high energy density (HED) foods. Participants receive breakfast, lunch and snack items engineered to have LPD and HED.
  Arms: Low physical and high energy density
Other: HPD+HED — High physical density (HPD) + high energy density (HED) foods. Participants receive breakfast, lunch and snack items engineered to have HPD and HED.
  Arms: High physical and energy density

SUMMARY:
As individuals tend to eat a constant weight or volume of food, manipulating physical and energy densities generally results in changes in energy intake without affecting subjective appetite sensations. However, relatively few studies have directly studied the interaction between physical and energy density manipulation. This study will determine the effects of foods that systematically vary in physical and energy density on ad libitum energy intake and subjective appetite ratings. Secondary outcomes will include gastrointestinal discomfort, fatigue and acceptability.

DETAILED DESCRIPTION:
A historical challenge for military personnel operating in austere, remote environments is the ability to pack and carry enough food to sustain their operational and nutritional needs. To address this challenge and meet Army modernization requirements, US Army ration developers are developing a new ration to provide a lightweight, low volume, energy dense daily combat assault ration. The ration will use novel food processing techniques that remove air and water to reduce volume and increase physical density (g/cc) and will provide a high relative fat content to increase energy density (kcal/g or kcal/cc). As individuals tend to eat a constant weight or volume of food, manipulating physical and energy densities generally results in changes in energy intake without affecting subjective appetite sensations. However, relatively few studies have studied the independent effects on appetite and energy intake of increasing physical and energy densities of foods to the extent being targeted by the new ration, and none has directly studied the interaction between physical and energy density manipulation. This study will address that gap by determining the effects of foods that systematically vary in physical and energy density on ad libitum energy intake and subjective appetite ratings. Secondary outcomes will include gastrointestinal discomfort, fatigue and acceptability. Using a randomized, crossover design consisting of four separate phases, 20 participants will be provided with a standard base diet and experimental foods in which physical and energy density are systematically varied using different levels of mechanical compression and aeration, and different proportions of fat and carbohydrate, respectively. Consumption of the experimental foods at each of the physical and energy density combinations will be compulsory for 1 day while intake of the standard diet will be ad libitum. Total energy and macronutrient intake will be measured by collecting uneaten food items. Additionally, perceived appetite, gastrointestinal symptoms, fatigue and acceptability of the experimental food products will be measured by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≤ 30.0 kg/m2
* Willing to abstain from alcohol for 24 hours prior to and during days 1-2 of each study phase.
* Willing to abstain from strenuous exercise for 24 hours prior to and during days 1-2 of each study phase.
* Willing to abstain from a vegetarian/vegan diet or other highly restrictive diet (e.g., ketogenic diet, very high protein diet, Paleo diet) for two weeks prior to and throughout the study.
* Willing to maintain body weight throughout study.
* Willing to maintain usual diet (if not a restrictive diet), physical activity (aside from strenuous exercise limitation for 24 hours prior to and days 1-2 of each study phase) and nicotine use throughout study.
* Willing to abstain from dietary supplements (e.g., metabolism boosters, appetite suppressants, weight loss aids) impacting appetite or metabolism (as determined by study PI) throughout the study.
* Eats 3 meals per day at least 5 days/wk

Exclusion Criteria:

* Pregnant or lactating.
* Taking prescription medications, other than a contraceptive, known to affect appetite, digestion and/or metabolism (e.g., anti-diabetic agents) (unless approved by study PI)
* Any chronic medical condition that limits food intake or alters metabolism, appetite or digestive physiology (e.g., gastric bypass, gastrointestinal disease, dysphagia, diabetes).
* Allergies and intolerances (e.g. gluten, dairy, nuts), unwillingness or inability to eat provided foods and beverages.
* Score of ≥13 on the restraint scale or ≥9 on the disinhibition scale of the Eating Inventory
* Weight gain or loss of >5 lbs in the 2 weeks prior to study participation.
* Not willing or unable to adhere to all study procedures and restrictions.

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Total energy intake | Day 1 of each study arm.
  Total energy intake from provided diet measured by weighing provided and uneaten foods.

SECONDARY OUTCOMES:
Carbohydrate intake | Days 1 and 2 of each study arm
  Total carbohydrate intake from provided and self-selected diet measured by weighing provided and uneaten foods, and food records.
Protein intake | Days 1 and 2 of each study arm
  Total protein intake from provided and self-selected diet measured by weighing provided and uneaten foods, and food records.
Fat intake | Days 1 and 2 of each study arm
  Total fat intake from provided and self-selected diet measured by weighing provided and uneaten foods, and food records.
Self reported energy intake | Day 2 of each study arm
  Energy intake from self-selected diet measured by food records.
Appetite | Immediately before, immediately after and 15 min after breakfast, lunch and afternoon snack on day 1 of each study arm
  Hunger, fullness, desire to eat and prospective consumption measured by 100mm visual analog scale. Range is 0 to 100, with higher scores indicating greater hunger/fullness/desire/prospective consumption.
Fatigue | Immediately before, immediately after and 15 min after breakfast, lunch and afternoon snack on day 1 of each study arm
  Level of fatigue measured by integer scale ranging from 0 (not tired) to 10 (total exhaustion)
Gastrointestinal symptoms | Immediately before, immediately after and 15 min after breakfast, lunch and afternoon snack on day 1 of each study arm
  Heartburn, bloating, abdominal pain, urge to vomit, nausea, gas, urge to defecate, overall gastrointestinal discomfort measured by 100mm visual analog scale. Range 0 (none) to 100 (extremely severe).
Acceptability | At breakfast, lunch and afternoon snack on day 1 of each study arm
  Appearance, odor, flavor, texture, and overall acceptability of experimental foods rated on scale ranging from 1 (dislike extremely) to 9 (like extremely).

CONTACTS AND LOCATIONS:
Overall Officials: J. Philip Karl, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05408390/ICF_000.pdf